CLINICAL TRIAL: NCT03523494
Title: Feasibility of Lymph Edema-induced Reticulation Subtraction Based on Computerized Tomography.
Status: Completed | Type: Observational
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Hwang, Associate professor, PhD and MD, Ulsan University Hospital
Other Study IDs: chhwang9
Record Dates: First submitted 2018-04-17; First posted 2018-05-14 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Lymphedema; Secondary Lymphedema; CT
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal limb: Normal
- Abnormal limb: Lymph Edema

SUMMARY:
Development of lympho-proliferation reticulation quantification using CT.

DETAILED DESCRIPTION:
It is known that fibrosis of the subcutaneous soft tissue progresses over time in the lymph edema, and this change progresses to reticulation pattern.

Authors will develop a digital subtraction technique for the extraction of lympho-proliferative reticulation using the Housfield unit of non-reticulation structure (bones, muscles, tendons, vessels, nerves) in the axial image of CT.

Based on the medical records, authors will develop an early diagnosing tool by checking the correlation of the values derived the new technique with circumference, multi-frequency bio-electric impedance analysis, ISO sub-stage, and lymphascintigraphy, and qualify the cut-off values showing high sensitivity and specificity through the receiver operating characteristics (ROC) curve analyses.

ELIGIBILITY:
Inclusion Criteria:

* In- and out-patients who was diagnosed a secondary lymphoma and undertook CT on their limbs

Exclusion Criteria:

* Primary lymph edema (congenital lymph edema, lymph edema precox, lymph edema tarda)
* Lymph edema simultaneously involving both limbs
* Patients who undertook implantation of electrical devices such as cardic pacemakers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In- and out-patients who was diagnosed a secondary lymphoma and undertook CT on their limbs
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Reticulation Ratio from Computerized Tomography | 1 week
  calculated value of reticulation

SECONDARY OUTCOMES:
Multi-frequency bio-electric impedance analysis | 1 week
  comparative ratio using 1KHz

OTHER OUTCOMES:
International Society of Lymphology stage | 1 week
  stage Ia, Ib, IIa, IIb, IIIa, and IIIb
lymphascintigraphy stage | 1 week
  Normal: 1; delayed flow, but visible axillary lymph or inguinal lymph node: 2; , invisible axillary lymph or inguinal lymph node: 3: visible dermal backflow: 4
circumference between normal and involved limbs | 1 week
  5cm above and below mid-antecubital or mid-popliteal fossa

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Hwang, M.D., Ph.D., Study Director — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koo KI, Ko MH, Lee Y, Son HW, Lee S, Hwang CH. Comparison of a novel algorithm quantitatively estimating epifascial fibrosis in three-dimensional computed tomography images to other clinical lymphedema grading methods. PLoS One. 2019 Dec 10;14(12):e0224457. doi: 10.1371/journal.pone.0224457. eCollection 2019. PMID 31821335